CLINICAL TRIAL: NCT04229901
Title: Randomized, Placebo-controlled, Double Blind, Multi-centre Phase IIb Study to Evaluate the Efficacy and Safety of HepaStem in Patients With Acute on Chronic Liver Failure (ACLF
Brief Title: Study to Evaluate the Efficacy and Safety of HepaStem in Patients With Acute on Chronic Liver Failure (ACLF)
Acronym: DHELIVER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Cellaion SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEP102
Record Dates: First submitted 2020-01-06; First posted 2020-01-18 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Acute on Chronic Liver Failure
Keywords: ACLF; Hepastem; HALPC
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HepaStem (Experimental): Patients in the HepaStem arm will receive 2 infusions of HepaStem (i.v) at 1.0 million of cells/kg of total body weight (7 day interval)
  Interventions: Drug: HepaStem
- Placebo (Placebo Comparator): Patients in the placebo arm will receive 2 infusions of placebo (i.v) (7 day interval)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HepaStem — HepaStem will be administered as an intravenous (IV) infusion
  Arms: HepaStem
Drug: Placebo — Placebo will be administered as an intravenous (IV) infusion
  Arms: Placebo

SUMMARY:
This is an interventional, double blind, randomized (2:1), and placebo-controlled study of 2 infusions of a 1 dose regimen of HepaStem in patients recently diagnosed (≤1 week) with ACLF grade 1 or 2 on top of Standard of Care (SoC), and for whom the diagnosis is not resolved on the day of infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Are adults aged between 18 and 75 years old.
2. Have an initial diagnosis of ACLF at the investigational site.
3. Have ACLF grade 1 or 2 according to the EASL-CLIF Consortium definition.
4. Have a total bilirubin ≥ 5 mg/dL.
5. Are able to read, understand and give written informed consent.

Main Exclusion Criteria:

1. Have a MELD-Na score > 35.
2. Have underlying cirrhosis due to biliary disease.
3. Have underlying cirrhosis due to autoimmune hepatitis.
4. Have active bleeding at a non-compressible site or at a compressible site that, in the opinion of the investigator, poses an unacceptable risk for the patient's participation in the study.
5. Have received treatment for bleeding complications during the current hospitalization and has a persistent high risk for re-bleeding that, in the opinion of the investigator, poses an unacceptable risk for the patient's participation in the study.
6. Have a complete portal vein thrombosis.
7. Have coagulation disturbances defined as:

   * fibrinogen < 80 mg/dL
   * platelets < 50 x 10³/mm³
8. Are requiring chronic dialysis therapy.
9. Have had a cerebrovascular, myocardial, limb arterial thrombotic event, or history for both thrombotic and hemorrhagic cerebrovascular events within 12 months prior to the Screening and not considered stabilized by the investigator.
10. Have a previous history of myocardial infarction and/or cardiac failure, with an ejection fraction rate (EFR) ≤ 40%.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Survival | Day 90
  Whether the patients are still alive will be recorded up to Day 90. Time and reason of death will be recorded.

SECONDARY OUTCOMES:
Liver transplant-free survival | Day 90
Transplant-free survival while free of ACLF | Day 90
Transplant-free survival with MELD-Na score < 15 | Day 90
Duration of overall hospitalization and hospitalization in ICU and non-ICU during the index hospitalization | up to Day 90

CONTACTS AND LOCATIONS:
Locations (47):
- Medical University Of Vienna, Vienna, Austria
- Belgium (7):
  - UZ Antwerpen, Antwerp
  - CHU Brugmann, Brussels
  - CHU Erasme, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - CHC MontLégia, Liège
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Bulgaria (5):
  - University Multiprofile Hospital for Active Treatment "Dr. Georgi Stranski", Pleven
  - UMHAT Medica, Rousse
  - Military Medical Academy, Sofia
  - UMHAT Sveta Anna, Sofia
  - UMHAT Tzarita Joanna, Sofia
- Aarhus University Hospital, Aarhus, Denmark
- Estonia (2):
  - North Estonia Regional Hospital, Tallinn
  - Lääne-Tallinna Keskhaigla AS, Tallinn
- France (11):
  - CHU Angers, Angers
  - Hopital Beaujon, Clichy
  - Assistance Publique Hopitaux De Paris, Créteil
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - Hospices Civils De Lyon, Lyon
  - Assistance Publique Hopitaux De Marseille, Marseille
  - CHU Montpellier, Montpellier
  - Assistance Publique-Hopitaux de Paris - Hopitaux Universitaires Pitie-Salpetriere, Paris
  - Les Hopitaux Universitaires De Strasbourg, Strasbourg
  - CHU De Toulouse, Toulouse
  - Hospital Paul Brousse, Villejuif
- Germany (3):
  - Medizinische Hochschule Hannover, Hanover
  - University Hospital Of Leipzig, Leipzig
  - University Hospital Of Ulm AöR, Ulm
- Italy (3):
  - Azienda Ospedaliera Ospedale Niguarda CA' Granda, Milan
  - Azienda Ospedaliera Universitaria Policlinico, Palermo
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Lietuvos Sveikatos Mokslų Universiteto Ligoninė Kauno Klinikos, Kaunas, Lithuania
- North Macedonia (2):
  - PHI General City Hospital "8mi Septemvri", Skopje
  - PHI University Clinic of Gastroenterohepatology, Skopje
- Poland (2):
  - Id Clinic, Mysłowice
  - Kliniczny Szpital Wojewódzki Nr 2 Im. Św. Jadwigi Królowej W Rzeszowie, Rzeszów
- F.D. Roosevelt University General Hospital Of Banská Bystrica, Banská Bystrica, Slovakia
- Spain (7):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - University Hospital Ramón Y Cajal, Madrid
  - Hospital Universitario Puerta De Hierro De Majadahonda, Majadahonda
  - Sabadell Hospital, Sabadell
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Unviersitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://cellaion.com/